CLINICAL TRIAL: NCT07314606
Title: Open-Label Multicentre Randomized Dietary Intervention Study in Pediatric Crohn's Disease Patients Initiating Anti-TNF Therapy
Brief Title: Combining Nutritional Therapy and Anti-TNFα Treatment in Pediatric Patients With Crohn's Disease
Acronym: DISPENSE-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kevan Jacobson, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H25-02014; GR034356 (Other Grant/Funding Number: Canadian IBD Research Consortium (CIRC))
Record Dates: First submitted 2025-09-29; First posted 2026-01-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD); IBD (Inflammatory Bowel Disease); IBD - Inflammatory Bowel Disease
Keywords: CDED; Exclusion Diet; Infliximab; Nutritional therapy; Pediatric; Diet Intervention
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFX + mCDED (Experimental): Participants will follow the modified Crohn's disease exclusion diet (mCDED) for 6 months, when initiating their infliximab therapy as part of their routine care
  Interventions: Other: IFX + mCDED
- IFX (No Intervention): Participants will initiate their infliximab therapy as part of their routine care

INTERVENTIONS:
Other: IFX + mCDED — modified Crohn's Disease Exclusion Diet (mCDED) ; Diet intervention
  Arms: IFX + mCDED

SUMMARY:
Children with Crohn's disease (CD), a type of Inflammatory Bowel Disease (IBD), often face serious health challenges, including poor growth, frequent hospital stays, and long-term medication use. Although biologic drugs like infliximab, an anti-TNFα (Tumor necrosis factor α) medication, have improved treatment, they don't work for everyone: many children still experience symptoms or disease flare-ups. Nutritional therapies, especially the Crohn's Disease Exclusion Diet (CDED), may help improve treatment outcomes. This study will assess whether starting CDED at the same time as infliximab leads to better responses to treatment. The goal of this study is to improve how well children respond to therapy, reduce drug exposure, and support better long-term health.

DETAILED DESCRIPTION:
This open-label, randomized, controlled interventional study will evaluate the effectiveness of combining nutritional therapy (modified Crohn's Disease Exclusion Diet; mCDED) with infliximab (IFX) in pediatric patients with luminal Crohn's disease (CD), compared to IFX alone.

The investigators hypothesize that initiating mCDED at the start of IFX therapy will enhance clinical response by the time the first IFX maintenance dose is given (week 12), and increase clinical and biochemical remission rates at 1 year (week 52).

Participation will last up to 16 months and includes a pre-randomization phase of up to 4 months (for baseline sample and data collection), and 12 months of intervention. After randomization (T0), participants assigned to the intervention arm will follow a standardized IFX infusion schedule and begin the mCDED with the support of a dietitian. Participants in the control arm will follow the same IFX schedule and meet with a dietitian who will review their usual eating habits, but they will not be asked to follow any dietary advice.

A total of 140 pediatric CD patients (70 per arm) will be recruited from the lead site (Vancouver) and 7-9 additional participating sites (Montreal, Ottawa, Toronto, Halifax, Calgary, Edmonton, London, Hamilton) within the Canadian Children Inflammatory Bowel Disease Network (CIDsCaNN).

The following samples and data will be collected:

1. 3-day diet record (3DDR) - Completed by both arms at weeks 1, 12, 24 and 52 to assess dietary intake differences and dietary adherence to mCDED.
2. 24-hour diet recall - Conducted by a dietitian to assess dietary adequacy of both groups at weeks 1, 2 (for intervention group only), 6, 12, and 24.
3. CDED diet habits questionnaire - Completed by both groups at weeks 1 and 52 to assess how their diet aligns with the mCDED and to evaluate any changes in dietary habits.
4. CDED adherence questionnaire - Completed by the intervention group only at weeks 2, 6, 12, and 24.
5. KIDMED questionnaire (Mediterranean Diet Quality Index in children) - Completed by both groups at weeks 1 and 52 to assess adherence to a healthy diet and good dietary habits.

7) Paediatric Yorkhill Malnutrition Score (PYMS) - At pre-randomization assessment, weeks 24 and 52, to assess malnutrition.

8) Clinical and Biochemical Data - Weighted paediatric Crohn's disease activity index (wPCDAI), physician global assessment (PGA), C-reactive protein (CRP), ESR (Erythrocyte Sedimentation Rate), Fecal calprotectin (FCP) and hematological data (Complete Blood Count [CBC]) collected at pre-randomization assessment, weeks 1, 6, 12, 24 and 52.

9) Anthropometric data (body mass index [BMI], growth velocity) - Assessed over study at pre-randomization assessment, weeks 1, 2, 6, 12, 24, 36 and 52.

10) Nutritional status (Albumin, Ferritin, B12, Vitamin D levels) - Measured in blood at weeks 1, 6, 12, 24 and 52 11) IFX trough levels - Measured in blood at weeks 6, 12, 24 and 52. 12) Optional blood sample - Participants will have the option to provide a blood sample during the pre-randomization assessment for genetic testing to investigate genetic variants that may influence response to IFX, including but not limited to HLADQA1*05 (major histocompatibility complex, class II, DQ alpha 1).

13) Magnetic Resonance Elastography (MRE) - Performed at Baseline (within 4 months prior to randomization and starting therapy) and at week 52 (±4 weeks) and/or when clinically indicated to assess disease activity.

14) Intestinal ultrasound (IUS) - Performed at Baseline (T-2, within 4 months prior to randomization and starting therapy), weeks 12 (±2 weeks), 24 (±4 weeks) and 52 (±4 weeks) to assess disease activity (transmural intestinal inflammation).

15) Colonoscopy - At Baseline (within 4 months prior to randomization and starting therapy) and at week 52 (±4 weeks) to assess disease activity (SES-CD; Simple endoscopic score for Crohn's disease). While not mandatory, it is highly encouraged. In the absence of a colonoscopy, a composite score will be generated. If a colonoscopy is performed, mucosal washes and intestinal biopsies will be collected for research purpose.

16) Fecal samples - Collected without preservatives by participants at weeks 1, 2, 6, 12, 24, and 52 for longitudinal microbiota analysis, in vitro microbiota culturing, and fecal transplantation into germ-free recipient mice.

17) IMPACT-III - Quality of life survey completed by all participants at weeks 1, 12 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe active luminal inflammatory (B1) pCD [wPCDAI > or = 40] ileal +/- colonic (L1, L2, L3), and in whom treating physician plans to start IFX
* OR Strong suspicion of moderate-severe active luminal inflammatory (B1) pCD ileal +/- colonic (L1, L2, L3), and in whom treating physician plans to start IFX
* Within 12-months of diagnosis (when starting IFX treatment)
* Naïve to a biologic therapy
* For patients with established disease who flare up: no response to dietary intervention or steroids within 4 weeks of commencement of these therapies.
* For newly diagnosed patients: no response to dietary intervention or steroids within 2 weeks of commencement of these therapies.
* Evidence of active inflammation: FCP level > 250 µg/g and/ or CRP > 5 mg/L or ESR > 20 mm/hr
* BMI between the 5th and 95th percentiles, adjusted for age and sex
* On steroids or EEN for less than 2 (or 4, for established disease) weeks
* Able and willing to follow dietary recommendations
* On stable dose of AZA or Methotrexate (MTX) at randomization
* Willing to enroll in the CIDsCaNN Network study

Exclusion Criteria:

* CDED, EEN, or steroids commenced more than 2 weeks prior to randomization
* Antibiotic use in the last 2 months (except short course < 1 week between 1-2 months) or laxative use within the past month (except for bowel prep for endoscopy pre commencement of anti-TNFα)
* Pre-, pro-, synbiotic supplements in the last month (food containing these products, e.g. yogurt, allowed)
* Strict vegetarians and vegans
* High risk of malnutrition as assessed by the Paediatric Yorkhill Malnutrition Score (PYMS)
* Other known GI disorders (except IBS), food intolerances or chronic diseases
* Bowel surgery prior the randomization
* Severe perianal disease (fistulizing or ulcerating), fibrostenotic (B2) or penetrating (B3) disease
* Currently on prednisone/prednisolone for > 2 weeks
* Pregnant or breastfeeding
* Participating in another study
* Inability to consent

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and biochemical response at the first infliximab (IFX) maintenance dose (week 12) in participants receiving mCDED alongside IFX compared with participants receiving IFX alone. | 12 weeks
  Clinical response: defined as mild or inactive clinical disease (at least a 17.5-points decrease in weighted paediatric Crohn's disease activity index (wPCDAI) from baseline, with a score < 40), physician global assessment (PGA) of inactive or mild disease activity, off steroids, continuation on the same anti-TNFα dose, and remaining surgery-free.
  Biochemical response: Defined as at least a 50% decrease in fecal calprotectin (FCP) levels compared to baseline.
  wPCDAI ranges from 0 to 125, with higher scores indicating greater disease activity.
  PGA ranges from 0 to 10, with higher scores indicating greater disease activity.

SECONDARY OUTCOMES:
Steroid-free clinical and biochemical remission at week 12 in participants receiving mCDED alongside IFX compared with participants receiving IFX alone. | 12 weeks
  Steroid-free clinical remission (SFCR): defined as an inactive disease (wPCDAI <12.5), PGA of inactive disease, no steroid use in the preceding 28 days, continuation on IFX and remaining surgery-free.
  Biochemical remission: defined as a normalization of C-reactive protein (CRP) (< 5 mg/L) and Erythrocyte Sedimentation Rate (ESR) (< 15-20 mm/h, male & female respectively) if available, and FCP level < 250 µg/g.
  wPCDAI ranges from 0 to 125, with higher scores indicating greater disease activity.
  PGA ranges from 0 to 10, with higher scores indicating greater disease activity.
Steroid-free clinical and biochemical response at weeks 24 and 52 in participants receiving mCDED alongside IFX compared with participants receiving IFX alone. | 24 and 52 weeks
  Steroid-free clinical response: defined as mild or inactive clinical disease (at least a 17.5-points decrease in weighted paediatric Crohn's disease activity index (wPCDAI) from baseline, with a score < 40), physician global assessment (PGA) of inactive or mild disease activity, off steroids, continuation on the same anti-TNFα dose, and remaining surgery-free.
  Biochemical response: Defined as at least a 50% decrease in fecal calprotectin (FCP) levels compared to baseline.
  wPCDAI ranges from 0 to 125, with higher scores indicating greater disease activity.
  PGA ranges from 0 to 10, with higher scores indicating greater disease activity.
Proportion of participants achieving steroid-free clinical and biochemical remission at weeks 24 and 52 in participants receiving mCDED alongside IFX compared with participants receiving IFX alone. | weeks 24 and 52
  Steroid-free clinical remission (SFCR): defined as an inactive disease (wPCDAI <12.5), PGA of inactive disease, no steroid use in the preceding 28 days, continuation on IFX and remaining surgery-free.
  Biochemical remission: defined as a normalization of C-reactive protein (CRP) (< 5 mg/L) and Erythrocyte Sedimentation Rate (ESR) (< 15-20 mm/h, male & female respectively) if available, and FCP level < 250 µg/g.
  wPCDAI ranges from 0 to 125, with higher scores indicating greater disease activity.
  PGA ranges from 0 to 10, with higher scores indicating greater disease activity.
1-year composite score of clinical remission and biochemical remission in addition to meeting criteria for steroid-free clinical remission adjusted for week 12 IFX trough level. | Week 52
  1-year composite score remission: defined as the concurrent achievement of clinical remission and biochemical remission at the 12-month follow-up. This score will be adjusted by the IFX blood level (in µg/mL) measured at week 12.
  Steroid-free clinical remission (SFCR): defined as an inactive disease (wPCDAI <12.5), PGA of inactive disease, no steroid use in the preceding 28 days, continuation on IFX and remaining surgery-free.
  Biochemical remission: defined as a normalization of C-reactive protein (CRP) (< 5 mg/L) and Erythrocyte Sedimentation Rate (ESR) (< 15-20 mm/h) if available, and FCP level < 250 µg/g.
  1-year composite score: 0 = no remission
  1. = clinical or biochemical remission
  2. = clinical and biochemical remission
Endoscopic response and endoscopic remission at week 52 in participants receiving mCDED alongside infliximab (IFX) compared with participants receiving IFX alone. | Week 52
  Endoscopic response: defined as at least a 50% reduction from baseline in Simple endoscopic score for Crohn's disease (SES-CD), or for patients with isolated ileal disease and a baseline SES-CD of 4, at least a 2-point reduction from baseline.
  Endoscopic remission: defined as an SES-CD score lower or equal to 4, with at least a 2-point reduction from baseline and no sub-score > 1. Deep remission as per wPCDAI and endoscopic remission.
  SES-CD ranges from 0 to 56, with higher scores indicating greater disease activity.
Frequency of progression from inflammatory phenotype (B1) to complicated disease (B2, B3, or B2/B3) in participants receiving mCDED alongside IFX compared with participants receiving IFX alone. | Week 52
  Disease progression will be evaluated by assessing whether participants with an initial inflammatory phenotype (B1) develop a stricturing (B2), penetrating (B3), or mixed (B2/B3) phenotype during follow-up, based on the Montreal classification. Progression will be confirmed through cross-sectional imaging (MRE, or IUS), colonoscopy, or surgical findings showing luminal narrowing, pre-stenotic dilation, or fistula/abscess formation. Imaging will be performed at baseline and as clinically indicated. The number of participants progressing from B1 to B2/B3 and time to first progression from B1 to B2/B3 will be recorded.
Long-term dietary habits in participants receiving dietary therapy, including consumption of ultra-processed foods (UPFs) and adherence to healthy dietary patterns. | Week 52
  Participants will fill out the KIDMED questionnaire at baseline and at week 52.
  The KIDMED score is a 16-item questionnaire used to assess a child or adolescent's adherence to the Mediterranean Diet (MD). The total score ranges from -4 to +12. Value of the KID-MED score: ≤3, very-low-quality diet; 4-7, need to improve the food pattern to adjust it to the Mediterranean one; ≥8, optimal Mediterranean diet.
Association between ongoing adherence to reduced ultra-processed food (UPF) consumption and long-term biologic response. | Week 52
  The relationship between KIDMED score and clinical and biochemical response or remission will be investigated.
  The KIDMED score is a 16-item questionnaire used to assess a child or adolescent's adherence to the Mediterranean Diet (MD). The total score ranges from -4 to +12. Value of the KID-MED score: ≤3, very-low-quality diet; 4-7, need to improve the food pattern to adjust it to the Mediterranean one; ≥8, optimal Mediterranean diet.
  Clinical response: defined as mild or inactive clinical disease (at least a 17.5-points decrease in weighted paediatric Crohn's disease activity index (wPCDAI) from baseline, with a score < 40), physician global assessment (PGA) of inactive or mild disease activity, off steroids, continuation on the same anti-TNFα dose, and remaining surgery-free.
  Biochemical response: Defined as at least a 50% decrease in fecal calprotectin (FCP) levels compared to baseline.
Microbial changes induced by the dietary intervention and their association with clinical and biochemical response. | Weeks 12, 24 and 52
  Microbial analyses that will be undertaken for each sample type are as follows:
  Stool:
  * Metagenomics (Shotgun sequencing, ITS sequencing for fungal analysis)
  * Metaproteomics and metabolomics (Host, microbial, and dietary protein analysis, microbial metabolite analysis)
  * Anaerobic culturing (Simulate gut environment, use dietary substrates to target key microbes)
  Biopsy specimens:
  * RNA-seq, transcriptomics (Gene expression profiling analysis, disease marker identification)
  * Metagenomics
  * Metaproteomics and metabolomics
  Intestinal washings:
  * Metagenomics
  * Metaproteomics and metabolomics
Association between baseline microbiome profiles and therapeutic outcomes at the first IFX maintenance dose (week 12) using compositional analyses and machine learning (ML) approaches. | Week 12
  Multi-modal integrative analysis will combine metagenomic, metaproteomic, and metabolomic data with diet (mCDED vs. regular diet), endoscopic and clinical scores (SES-CD, PCDAI), biochemical markers (FCP, ESR, CRP), quality of life, and anthropometric data. Univariate analyses will be performed to test associations between each quantitative measure of disease activity and each dataset (taxonomic and functional tables), identifying both positive and negative correlations. Sparse Partial Least Squares Discriminant Analysis (sPLS-DA; http://mixomics.org/) will be used for feature selection and dimensionality reduction to identify the most informative predictors. These features will then be used to train predictive models with Random Forest classifiers and artificial neural networks (ANN), providing complementary approaches for robust prediction. Model performance and generalizability will be evaluated using repeated cross-validation (20 × 5-fold).

CONTACTS AND LOCATIONS:
Overall Officials: Kevan Jacobson, MBBCh, FRCP, FRCPC, AGAF, CAGF, Principal Investigator — The University of British Columbia; Genelle Lunken, BSc, PhD, RD, Principal Investigator — The University of British Columbia
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared with researchers in the future; however, the specific details of the data sharing plan have not yet been finalized. Therefore, we are selecting "Undecided" at this time and will update the response to "Yes" once the strategy has been refined.